CLINICAL TRIAL: NCT02680054
Title: Investigation of Appropriate Timing of Additional Insulin Dosing for Fat and Protein in Children With Type 1 Diabetes Using Multiple Daily Injections
Brief Title: Additional Insulin for Fat and Protein in Children With Diabetes Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No eligible participants left to approach/ recruit
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Rachel Besser, Consultant in Paediatric Diabetes, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 114185; 2015-003666-85 (EudraCT Number)
Record Dates: First submitted 2016-02-04; First posted 2016-02-11 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (usual treatment) (Active Comparator): Insulin dose (insulin Aspart, NovoRapid) for the fat and protein in a high-fat, high-protein meal is given at the same time as the insulin for the carbohydrate content BEFORE the meal. The dose is calculated on an individual basis according to the usual insulin to carbohydrate ratio for that child.
  Interventions: Drug: Insulin, Asp(B28)-
- Arm 2 (Active Comparator): Insulin dose (insulin Aspart, NovoRapid) for the fat and protein in a high-fat, high-protein meal is given one hour after the meal. The dose is calculated on an individual basis according to the usual insulin to carbohydrate ratio for that child.
  Interventions: Drug: Insulin, Asp(B28)-
- Arm 3 (Active Comparator): Insulin dose (insulin Aspart, NovoRapid) for the fat and protein in a high-fat, high-protein meal is given two hours after the meal. The dose is calculated on an individual basis according to the usual insulin to carbohydrate ratio for that child.
  Interventions: Drug: Insulin, Asp(B28)-

INTERVENTIONS:
Drug: Insulin, Asp(B28)- — This insulin dose is sometimes given for fat and protein content of food in children using insulin pumps, in prolonged boluses. The investigators are replicating this in children using multiple insulin injections at various times related to the meal
  Other Names: NovoRapid

SUMMARY:
The aims of the study are to see if additional insulin doses for the fat and protein in a meal, given at different times, improve blood glucose levels and are safe and acceptable to children with Type 1 diabetes using multiple daily insulin injections.

DETAILED DESCRIPTION:
The study design is a repeated measures study involving the provision of a standard high protein/high fat evening test meal on 3 different evenings within a 7-day period in the same study subject. The children/adolescents will be instructed to give an insulin dose for the carbohydrate before the meal (calculated using their optimal insulin to carbohydrate (ICR) - 20%). In addition they will have an additional dose for the fat and protein content either before (together with the dose for the carbohydrate in the meal [control meal]), 1 hour after, or 2 hours after the meal. These will be carried out in a random order in each subject. Continuous glucose monitoring (CGM) will be carried out for the whole 7 day period. Questionnaires will assess the acceptability to young people and their parents of the extra insulin doses.

After an initial contact in the clinic, and provision of patient information leaflets, the research nurse or dietitian will telephone the patient and family after a week to answer any questions they may have about the study. If they are keen to participate, an appointment will be arranged for consent and to commence the study (Visit 1).

At Visit 1 the investigators will obtain informed consent and commence a week-long run-in period for participants to optimise insulin to carbohydrate ratio at the evening meal. During this week subjects will be requested to test capillary blood glucose (BG) levels at 7 points throughout the day (pre-meals, 2 hrs after meals and bed). They will be asked to eat a fat and protein free meal on one of these days. If necessary, adjustments to the insulin to carbohydrate ratio (ICR) or long-acting insulin doses will be made over the telephone by an experienced member of their clinical team. This is to decrease the likelihood of a correction bolus for a high BG level being required at the evening meal during the study week.

At the end of the run-in week, participants will then attend the outpatient clinic or day care ward research facility at the Oxford Children's Hospital or the Horton Hospital outpatient clinic in Banbury or the Royal Berkshire Hospital in Reading (Visit 2). At this visit, the subcutaneous glucose sensor will be inserted by the research nurse and children and young people and their families will be trained on its use prior to the study commencing. CGM records glucose levels every 5 minutes over 7 days and thus provides much more information than routine capillary BG testing. It also alarms to alert patients of high and low glucose levels. Children and young people will also record their BG levels from routine finger pricks, pre-prandially and before bed and on waking in the morning.

Also at Visit 2, the study dietitian will review BG readings and food diary from the previous week and optimise ICR doses of rapid acting insulin. This ratio will then be used to calculate insulin doses for the study meals. On three evenings over the next 7 days, the children will eat a standard high protein/high fat meal. The evenings will not be set, but will depend on the child and family schedule. The child and family will be able to choose which days during the study period on which they complete the study meals but will be advised to avoid days when the participant has undertaken lots of exercise, has had frequent hypoglycaemic episodes or has been unwell.

The standard meal will be a portion controlled gluten-free meal provided and delivered by Wiltshire Farm Foods consisting of a meat-based main course and dessert. These will be kept frozen until used by participants and prepared according to manufacturer instructions. These meals come in two sizes which allow portion sizes to be adjusted for different ages of child, but the proportions of fat, protein and carbohydrate will be kept constant for each child, and by definition the meals will be high in protein and high in fat.

Insulin doses with the standard meal will be given according to calculations carried out by the dietitian and administered in one of three ways.

The three evenings in random order will be as follows:

1. Insulin units based on ICR minus 20%, and fat/protein dose given together immediately before the meal [control meal].
2. Insulin units based on ICR minus 20%, given immediately before the meal plus extra insulin for fat/protein units given 1 hour after the meal.
3. Insulin units based on ICR minus 20% given immediately before the meal plus extra insulin for fat/protein units given 2 hours after the meal.

Full written instructions will be provided to the family for all aspects of the insulin dosing for the study meals. During the study on the standardised meal days children will be instructed not to eat any food after the meal during the evening, and not to correct any later BG levels unless they are dangerously high (BG over 16 mmol/l with ketones over 0.5 mmol/l). If BG levels go low at any time (BG less than 4 mmol/l) children will be instructed to treat the hypoglycaemia according to their usual management. This data will be analysed separately. Children and families will be asked to complete diaries during the trial week.

At the end of the study period (the day after the third meal), children will come back to the research facility or clinic for the end of study visit (visit 3). A research nurse or dietitian will remove the CGM sensor and download the data onto a secure laptop. Children and their families will then be asked to complete a short questionnaire about the acceptability of using the extra insulin doses, and their perceptions as to whether there were any beneficial or adverse effects.

The study dietitian will calculate standard outcomes from each patient's sensor download and pass on anonymously to the study statistician to analyse the data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 diabetes (for at least a year)
* On multiple daily insulin injections, including basal long-acting insulin and rapid-acting insulin before each meal.
* HbA1c < 75 mmol/mol (9.0%)
* Participant and/or parent/legal guardian willing and able to give informed consent for participation in the study.
* Family have a freezer in which to safely store the test meals.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* HbA1c greater than 75 mmol/mol (9.0%)
* Child unwilling to agree to second insulin injection at a meal-time
* Untreated coeliac disease or other concomitant condition likely to affect BG control
* Food allergies (other than controlled Coeliac Disease)
* Vegetarians, vegans or patients with religious dietary restrictions (as the standard meal contains meat)
* Participant taking any glucose-containing medication concurrently

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel E Besser, PhD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - Royal Berkshire Hospital, Reading, Berkshire
  - Oxford Children's Hospital, John Radcliffe Hospital, Oxford, Oxon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was closed before target could be reached due to exhaustion of eligible participants
Groups:
- All Study Participants: Insulin dose (insulin Aspart, NovoRapid) for the fat and protein in a high-fat, high-protein meal is given at the same time as the insulin for the carbohydrate content BEFORE the meal, then +1hr after, then +2hr after. The dose is calculated on an individual basis according to the usual insulin to carbohydrate ratio for that child.
  Insulin, Asp(B28)-: This insulin dose is sometimes given for fat and protein content of food in children using insulin pumps, in prolonged boluses. The investigators are replicating this in children using multiple insulin injections at various times related to the meal
Period: Overall Study
Arm/Group | All Study Participants
Started | 38
Completed | 27
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Insulin dose (insulin Aspart, NovoRapid) for the fat and protein in a high-fat, high-protein meal is given at the same time as the insulin for the carbohydrate content BEFORE the meal, then +1hr, then +2hr. The dose is calculated on an individual basis according to the usual insulin to carbohydrate ratio for that child.
  Insulin, Asp(B28)-: This insulin dose is sometimes given for fat and protein content of food in children using insulin pumps, in prolonged boluses. The investigators are replicating this in children using multiple insulin injections at various times related to the meal
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 27
Duration of T1 Diabetes [Mean (Full Range); unit: years] | 3.5 [1 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Peak Glucose Level Following Test Meal
Description: Glucose measured on the continuous subcutaneous glucose monitor
Time Frame: assessed up to 12 hours following the test meal
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Arm 1 (Usual Treatment) | Arm 2 | Arm 3
Number analyzed (Participants) | 27 | 27 | 27
mmol/l | 10.931 (0.951) | 11.491 (0.831) | 11.491 (0.863)

2. Primary Outcome: Peak Glucose Excursion From Baseline Following Test Meal
Description: Glucose measured on the continuous subcutaneous glucose monitor
Time Frame: assessed up to 12 hours following the test meal
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Arm 1 (Usual Treatment) | Arm 2 | Arm 3
Number analyzed (Participants) | 27 | 27 | 27
mmol/l | 1.864 (0.716) | 1.167 (0.72) | 2.459 (0.712)

3. Primary Outcome: Time of Peak Glucose Level Following Test Meal
Description: Glucose measured on the continuous subcutaneous glucose monitor
Time Frame: assessed up to 12 hours following the test meal
Measure: Mean (Standard Deviation); unit: Mins
Arm/Group | Arm 1 (Usual Treatment) | Arm 2 | Arm 3
Number analyzed (Participants) | 27 | 27 | 27
Mins | 82.34 (35.37) | 113.617 (30.922) | 95.106 (32.092)

4. Secondary Outcome: Number of Participants With Hypoglycaemia Events Following the Insulin Dosing
Description: All episodes of hypoglycaemia (BG less than 4 mmol/l) either on continuous glucose monitor or self-monitoring of BG
Time Frame: assessed up to 12 hours following the test meal
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Usual Treatment) | Arm 2 | Arm 3
Number analyzed (Participants) | 27 | 27 | 27
Participants | 14 | 14 | 16

5. Other Pre Specified Outcome: Acceptability of Giving Insulin at Different Times Related to Test Meal
Description: Would young people continue to give extra insulin injections for High Fat High Protein (HFHP) meals
Time Frame: questionnaires completed up to a week after the test meals
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 27
Participants | 11

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Arm 1 (Usual Treatment) | Arm 2 | Arm 3
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT02680054/Prot_SAP_000.pdf